CLINICAL TRIAL: NCT01122511
Title: Safety and Efficacy of Dexamethasone as Adjunctive Therapy to Ranibizumab in Subjects With Choroidal Neovascularization and Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to difficulties with patient recruitment.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206207-021
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Subfoveal Choroidal Neovascularization; Age-Related Maculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 700 ug dexamethasone and ranibizumab (Experimental): Intravitreal injection of 700 ug dexamethasone and ranibizumab into study eye
  Interventions: Drug: 700 ug dexamethasone; Biological: ranibizumab
- ranibizumab and sham (Active Comparator): Intravitreal injection of ranibizumab and Sham into study eye
  Interventions: Biological: ranibizumab; Other: sham

INTERVENTIONS:
Drug: 700 ug dexamethasone — Intravitreal injection of 700 ug dexamethasone into study eye
  Other Names: OZURDEX®
  Arms: 700 ug dexamethasone and ranibizumab
Biological: ranibizumab — Intravitreal injection of ranibizumab into study eye
  Other Names: Lucentis®
Other: sham — Sham needle-less injection administered in the study eye
  Arms: ranibizumab and sham

SUMMARY:
This study will evaluate the safety and efficacy of dexamethasone (OZURDEX®) as adjunctive therapy to ranibizumab (LUCENTIS®) compared with ranibizumab alone in the treatment of patients with choroidal neovascularization secondary to age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Received at least 2 and no more than 3 monthly Lucentis or Avastin injections
* Last Lucentis or Avastin was injected approximately 4 weeks prior to screening
* Visual acuity between 20/320 and 20/40

Exclusion Criteria:

* Active ocular infection
* Contraindication to pupil dilation in either eye
* Eye surgery including cataract surgery and/or laser of any type within 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- United States (2):
  - Fort Myers, Florida
  - Abilene, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone and Ranibizumab: Intravitreal injection of 700 μg dexamethasone and ranibizumab into study eye.
Period: Overall Study
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Number; unit: Participants]
  Between 50 and 80 years | 1 | 0 | 1
  >=80 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 12
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Month 12
Population: No participants reached the 12 month time-point. Efficacy analyses were not performed.
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Percentage of Patients Having 15 or More Letter Improvement From Baseline in Best Corrected Visual Acuity at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: No participants reached the 12 month time-point. Efficacy analyses were not performed.
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness at Month 12 as Measured by Optical Coherence Tomography
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed on the study eye after pupil dilation at baseline and Month 12.
Time Frame: Baseline, Month 12
Population: No participants reached the 12 month time-point. Efficacy analyses were not performed.
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Area Leakage of Choroidal Neovascularization at Month 12 as Measured by Fluorescein Angiography
Description: Fluorescein angiography (FA) is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. FA was performed on the study eye after dilation at baseline and Week 12.
Time Frame: Baseline, Month 12
Population: No participants reached the 12 month time-point. Efficacy analyses were not performed.
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Dexamethasone and Ranibizumab | Ranibizumab and Sham
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone and Ranibizumab (N=2) | Ranibizumab and Sham (N=2)
Tooth Disorder (Gastrointestinal disorders) | 1 | 0
Retinal oedema (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulties with patient recruitment. No participants reached the 12 month time-point. Efficacy analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.